CLINICAL TRIAL: NCT00005660
Title: The Evaluation of Oral Acitretin in the Treatment of Psoriasis, Cutaneous Disorders of Keratinization, Multiple Basal Cell Carcinomas and Other Retinoid Responsive Diseases
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 770172; 77-C-0172; NCT00020956 (obsolete NCT alias)
Record Dates: First submitted 2000-05-12; First posted 2000-05-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-11

CONDITIONS: Basal Cell Carcinoma; Keratosis Palmaris et Plantaris; Psoriasis
Keywords: Hypertriglyceridemia; Teratogenicity; Ichthyosis; Darier's Disease; Retinoids; Skin; Psoriasis; Basal cell carcinoma; Skin Cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Keratoderma, Palmoplantar; Psoriasis; Hypertriglyceridemia; Teratogenesis; Ichthyosis; Darier Disease; Skin Neoplasms

SUMMARY:
This is a continuing study which evaluates the long-term safety and efficacy of oral acitretin in an open manner in the treatment of psoriasis, cutaneous disorders of keratinization, multiple basal cell carcinomas and other retinoid responsive diseases.

DETAILED DESCRIPTION:
This is a continuing study which evaluates the long-term safety and efficacy of oral acitretin in an open manner in the treatment of psoriasis, cutaneous disorders of keratinization, multiple basal cell carcinomas and other retinoid responsive diseases.

ELIGIBILITY:
Patients with widespread involvement (e.g. psoriasis patients with 10 percent or more of body surface area involved) or with severe, recalcitrant localized involvement with a cutaneous disorder (e.g. keratoderma palmaris et plantaris).

Patients (and parents of patients who are less than 18 years old) must be advised of presently available alternative forms of therapy.

Patient must be available for and agreeable to regular follow up examinations in the clinic for clinical evaluation, blood tests, diagnostic x-rays and possibly skin biopsies.

The patient (and parent, guardian, or surrogate where appropriate) must give written informed consent after protocol, including its limitations and risks, are thoroughly discussed with the patients (and parents).

Patients who have multiple skin cancers because of xeroderma pigmentosum (XP).

No patients with persistently abnormal (SGOT or SGPT greater than 3 times the upper limit of normal) liver function tests.

No patients with persistent pre-treatment hypertriglyceridemia (greater than 300 mg/dl).

No patients with persistently abnormal (creatinine greater than 3 times the upper limit of normal) renal function tests.

No patients with presence of a significant neurological, musculoskeletal or other internal medical disorder which may be aggravated by the addition of retinoid therapy.

Patient must not be pregnant or anticipate such an event. Because of the long-term storage of etretinate, a known teratogen, fertile women who may be treated in this protocol, must have skin disease that is severe and recalcitrant to all other standard modalities. These women must also use an effective form of contraception (oral contraceptives or an intrauterine device) while on treatment and at least for 3 years post treatment.

No patients with chronic intake of excessive dietary vitamin A (more than 25,000 iu/day).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 1977-10; Study Completion 2001-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States